CLINICAL TRIAL: NCT04530266
Title: Reliability of Measuring Walking-related Performance Fatigability Using Six Minute Walk Test in Persons With Knee Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Foundation University Islamabad (Other)
Collaborators: Hasselt University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: FUI/CTR/2020/6
Record Dates: First submitted 2020-08-25; First posted 2020-08-28 (Actual); Last update posted 2020-08-28 (Actual); Status verified 2020-08

CONDITIONS: Osteoarthritis; Osteoarthritis, Knee
Keywords: osteoarthritis; six minute walk test; reliability; fatigue; fatigability
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Fatigue | interventions — Walk Test

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Persons with knee osteoarthritis (Active Comparator)
  Interventions: Diagnostic Test: Six minute walk test
- Healthy controls (Placebo Comparator)
  Interventions: Diagnostic Test: Six minute walk test

INTERVENTIONS:
Diagnostic Test: Six minute walk test — Assessment of walking related performance fatigability using six minute walk test

SUMMARY:
Evidence has shown that knee osteoarthritis causes an increase in base of support and a decrease in stride length and gait velocity which results in an increase in energy expenditure during walking. This increase in energy cost of walking is suggested to result in walking related performance fatigability. However, fatigue is not commonly considered in the clinical settings in term of neither assessment nor management of knee osteoarthritis. One common tool used to evaluate walking relate performance is six minute walk test and the purpose of this study is to determine the reliability of using six minute walk test to determine walking related performance fatigability in persons with knee osteoarthritis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-70 years
* Knee OA with history not less than three months.
* Radiological evidences of grade III or less on Kellgren classification.
* Knee pain on VNRS no more than 8/10.

Exclusion Criteria:

* Neuromuscular conditions that may lead to fatigue such as multiple Sclerosis
* Signs of serious pathology (e.g., malignancy, inflammatory disorder, infection).
* History of trauma or fractures in lower extremity.
* Signs of lumbar radiculopathy or myelopathy.
* History of knee surgery or replacement.
* Patients on intra-articular steroid therapy within two months before the commencement of the study.
* Impaired skin sensation and renal function.

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2020-08-28 (Estimated); Primary Completion 2020-12-28 (Estimated); Study Completion 2020-12-28 (Estimated)

PRIMARY OUTCOMES:
Assessment of walking related performance fatigability using six minute walk test | Day 1
Assessment of walking related performance fatigability using six minute walk test | Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Osama, PhD*, Principal Investigator — Foundation University Islamabad
Locations (1):
- Foundation University Institute of Rehabilitation Sciences., Islamabad, Federal, Pakistan

IPD SHARING:
Plan to Share IPD: No